CLINICAL TRIAL: NCT02004795
Title: A Phase I/II Trial of Boron Neutron Capture Therapy (BNCT) Combined With Image-guided Intensity Modulated Radiotherapy (IG-IMRT) for Locally Recurrent Head and Neck Cancer
Brief Title: BNCT and IG-IMRT for Recurrent Head and Neck Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Tsing Hua University,Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-06-016A
Record Dates: First submitted 2013-11-11; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-11

CONDITIONS: Head and Neck Cancer; Recurrence
Keywords: Boron Neutron Capture Therapy; Image-guided intensity modulation radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence | interventions — Boron Neutron Capture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BNCT+ IG-IMRT (Experimental): single arm
  Interventions: Radiation: BNCT + IG-IMRT

INTERVENTIONS:
Radiation: BNCT + IG-IMRT — Single faction of BNCT (20 Gy) plus IG-IMRT (40 Gy/20 fractions)

SUMMARY:
This is a boron neutron capture therapy (BNCT) combined with image-guided intensity modulation radiotherapy (IG-IMRT) for patients with previously irradiated and locally recurrent head and neck cancer. The primary end points are treatment toxicities and response rate. The secondary endpoints are time to tumor progression, progression-free survival, overall survival and change quality of life.

Head and neck(H & N) carcinomas that recur locally after conventional irradiation pose a therapeutic challenge. Boron neutron capture therapy (BNCT) is based on the nuclear capture reaction that occurs when non-radioactive boron is irradiated with neutrons of thermal energy to yield high energy alpha particles and recoiling lithium nuclei. The effect of alpha and 7Li is primarily limited to boron-containing cells. Preferential uptake of boron into cancerous tissue is achieved using boron carriers such as a derivative of phenylalanine, boronophenylalanine (BPA). After administration of BPA by intravenous infusion, the tumor site is irradiated with neutrons, the source of which is currently a nuclear reactor, like the Tsing Hua Open-Pool Reactor (THOR), a 2MW research reactor at National Tsing Hua University (NTHU) in Taiwan. Since it is a target radiotherapy, low complication rate after BNCT can be obtained. However, further local recurrence after BNCT for recurrent H & N cancer was reported in several publications.

Image-guided radiation therapy (IGRT) is the process of frequent two and three-dimensional imaging, during a course of radiation treatment, used to direct radiation therapy utilizing the imaging coordinates of the approved radiation treatment plan. IGRT such as Cone-Beam CT (CBCT) using an On-Board Imager (OBI) enhance delivery and further improve outcomes as the treatments create a higher level of precision. By combining BNCT and IG-IMRT, we expect to procure high control rate of recurrent H & N cancer with acceptable toxicity. This study will be the first BNCT plus IG-IMRT trial to treat head and neck cancer in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* For BNCT:

  1. Patients with locoregionally recurrent, histologically proved malignancy of the head and neck, including primary sites of oral cavity, oropharynx, hypopharynx, nasopharynx, paranasal sinus, nasal cavity, the orbit, thyroid and larynx. Pathology types like melanoma and sarcoma are also included.
  2. Prior conventional radiotherapy administered has been given for the disease (except melanoma).
  3. Bi-dimensionally measurable disease by MRI and/or CT scan and ≦ 12 cm in largest dimension.
  4. Age greater than 18 years and < 80 years, ECOG performance status ≦ 2
  5. WBC > 2.5 x109/L, neutrophil count >1.0 x109/L, platelet count >75x109/L, serum creatinine <1.25xULN.
  6. Informed consent signed.
  7. Tumor/normal tissue (T/N) ratio≧2.5 by BPA-PET scan.
* For IG-IMRT:

  1. ECOG performance status ≦ 2
  2. No evidence of disease progression by physical examination or CT simulation.
  3. Nutrition support (feeding tube and/or IV fluid) already given for dysphagia, if present.
  4. Severity of mucositis and radiation dermatitis improved or downgrading, compared with those found in the 2nd or 3rd week after BNCT.

Exclusion Criteria:

* For BNCT:

  1. Lymphoma or other tumor type that is expected to respond to cancer chemotherapy or to a dose of conventional radiation therapy that can be safely given.
  2. Patients who have an effective standard treatment option available.
  3. Distant metastasis outside of the head and neck region.
  4. Expecting life less than 3 months.
  5. A time interval less than 6 months from previous radiation therapy.
  6. Prior high-dose radiotherapy (Biological Effective Dose> 70 Gy/35 fractions) has been given for the present recurrent site within one year.
  7. Patients who had radiation myelitis or radiation necrosis of the brain/brain stem
  8. Time to recurrence from completion of prior surgery less than 6 months.
  9. Concurrent systemic cancer treatment including chemotherapy or target therapy (including cetuximab or EGFR oral tyrosine kinase inhibitor).
  10. Severe congestive heart failure or renal failure.
  11. Pregnancy
  12. Restless patients who were unable to lie or sit in a cast for 30-60 min.
  13. A cardiac pace-maker or an unremovable metal implant present in the head and neck region that will interfere with MRI-based dose-planning or tumor response evaluation.
* For IG-IMRT:

  1. Any grade IV toxicity after BNCT.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
treatment toxicities | two years after combined treatment
  To evaluate both acute and late toxicities after combined BNCT and IG-IMRT
response rate | Three months after combined treatment
  including complete and partial response rate after BNCT+IG-IMRT

SECONDARY OUTCOMES:
Time to tumor progression | two years
  defined from the date of BNCT to the date of tumor progression by clinical evaluation.
Progression-free survival | two years
  calculated from the date of BNCT to the date of cancer progression either locally or distally or to death

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan